CLINICAL TRIAL: NCT06651853
Title: The Efficacy and Safety of Large Fraction Radiation Therapy Combined With Lenalidomide, and Glofitamab Monoclonal Antibody in the Treatment of Refractory Relapsed Diffuse Large B-cell Lymphoma Patients
Brief Title: Large Fraction Radiation Therapy Combined With Lenalidomide, and Glofitamab in Refractory Relapsed DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Zhijuan Lin, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-13
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-cell Lymphoma; Relapsed and Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Lenalidomide; glofitamab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Large fraction radiation therapy plus GM-CSF, Lenalidomide, and Glofitamab
  Interventions: Drug: Large fraction radiotherapy in combined with GM-CSF, Lenalidomide, and Glofitamab

INTERVENTIONS:
Drug: Large fraction radiotherapy in combined with GM-CSF, Lenalidomide, and Glofitamab — Large fraction radiotherapy is administered at 5Gy/day for 3 days, with one to two courses carried out on a single target lesion as determined by the investigator. Granulocyte-macrophage colony-stimulating factor (GM-CSF) is administered at 400µg per day for 3 days starting on the first day after the end of radiotherapy. Lenalidomide is administered at 25mg per day for 14 days starting on the first day after the end of radiotherapy. Glofitamab is administered starting on the 7th day after the end of radiotherapy.
  For cycles 2-6, each cycle is 21 days. GM-CSF is administered at 400µg per day for 3 days starting on the first day of each cycle. Glofitamab is administered at 30mg on the 4th day of each cycle. Lenalidomide is administered at 25mg per day for 14 days starting on the first day. Treatment consists of 6 cycles or until disease progression, death, intolerable toxicity, withdrawal of informed consent.

SUMMARY:
To prospectively evaluate the efficacy and safety of large fraction radiation therapy combined with granulocyte-macrophage colony-stimulating factor, lenalidomide, and glofitamab monoclonal antibody in the treatment of refractory relapsed diffuse large B-cell lymphoma patients

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any trial-related procedures are implemented.
2. Participants must be aged 18 or older, of any gender, with an expected survival period of more than 3 months.
3. ECOG PS score must be between 0-3.
4. Participants must have histopathologically confirmed diffuse large B-cell lymphoma.
5. Patients who have failed first-line standard treatment (patients with relapsed disease < 12 months or primary refractory disease, or relapsed disease > 12 months but are transplant-ineligible after 1 line of systemic therapy, or relapsed disease after 2+ lines of therapy). Participants with central nervous system metastasis can be included.
6. Participants must not have received bispecific antibody therapy in the past.
7. B-cell non-Hodgkin's lymphoma must have at least one measurable lesion according to RECIST1.1 criteria.
8. Participants must have sufficient organ function, meeting the following:

   laboratory criteria: (1) Total bilirubin ≤1.5× upper limit of normal (ULN); (2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× ULN; (3) Blood creatinine ≤1.5× ULN and creatinine clearance rate (calculated using the Cockcroft-Gault formula) ≥60 ml/min; (4) Good coagulation function, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN.
9. For women of childbearing potential, a urine or serum pregnancy test must be conducted within 3 days before the first administration of the study drug (Day 1 of Cycle 1) and the results must be negative. If the results of the urine pregnancy test cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing women are defined as those who have been menopausal for at least 1 year, or who have undergone surgical sterilization or hysterectomy.
10. If there is a risk of pregnancy, all participants (both male and female) must use contraception with an annual failure rate of less than 1% throughout the treatment period and for 120 days after the last administration of the study drug (or 180 days after the last chemotherapy administration).

Exclusion Criteria:

1. B-cell non-Hodgkin's lymphoma with loss of CD20 expression.
2. Acute or chronic active Hepatitis B or C infection, Hepatitis B virus (HBV) DNA>2000IU/ml or 104 copies/ml; Hepatitis C virus (HCV) RNA>103 copies/ml; simultaneous positivity for Hepatitis B surface antigen (HbsAg) and anti-HCV antibody.
3. Participants have received anti-hematologic malignancy treatment within 2 weeks before the start of treatment or within 5 half-lives of the drug, whichever is longer.
4. Bone marrow insufficiency defined by platelet count <30 x 109/L or absolute neutrophil count <1.0 x 109/L.
5. Participants with clinically significant pulmonary disease, including (1) participants with chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of the predicted normal value. Note that participants suspected of having COPD need to undergo an FEV1 test, and if FEV1<50% of the predicted normal value, the participant must be excluded. (2) Participants with moderate or severe persistent asthma in the past 2 years, or currently have any category of uncontrolled asthma. (Note that participants currently with controlled intermittent asthma or controlled mild persistent asthma can participate in this study).
6. Uncontrolled hypertension, with systolic blood pressure >150mmHg or diastolic blood pressure >90mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
7. Symptomatic congestive heart failure (New York Heart Association class II-IV). Symptomatic or poorly controlled arrhythmias. History of congenital long QT syndrome or a corrected QTc >500ms (calculated using the Fridericia method) at screening.
8. Large fraction radiation therapy received within 4 weeks prior to the first treatment. For patients who received radiation therapy more than 4 weeks before the first treatment, all the following conditions must be met to be included: there are currently no radiation-related toxic reactions, no need to take glucocorticoids, excluding radiation pneumonia, radiation hepatitis, radiation enteritis, etc.
9. Patients who have difficulty swallowing oral medications.
10. Past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function, and other lung diseases.
11. Human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive), known syphilis infection.
12. Presence of unhealed wounds, fractures, gastric and duodenal ulcers, persistent fecal occult blood positivity, ulcerative colitis, etc., or other conditions that the investigator determines may cause gastrointestinal bleeding or perforation.
13. Active or poorly controlled severe infection. Severe infection within 4 weeks before the first administration, including but not limited to hospitalization for complications of infection, sepsis, or severe pneumonia.
14. Major surgical treatment or significant traumatic injury received within 4 weeks before the first administration.
15. Traditional Chinese medicine with anti-tumor indications received within 2 weeks before the first administration.
16. Known allergy to any component of bispecific antibodies or GM-CSF formulations.
17. Treatment in another clinical trial within 4 weeks before the first administration.
18. Pregnant or breastfeeding female patients.
19. Presence of any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; participants who need bronchodilators for medical intervention for asthma cannot be included); but the following patients are allowed to participate: vitiligo, psoriasis, alopecia, well-controlled type I diabetes that does not require systemic treatment, and hypothyroidism with normal thyroid function through replacement therapy.
20. Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may lead to the following results: increase the risk associated with study participation or administration of the study drug, or interfere with the interpretation of study results, and according to the investigator's judgment, the patient is deemed ineligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
CR | Up to 36 months
  Complete remission rate, according to Lugano 2014 criteria.

SECONDARY OUTCOMES:
ORR | Up to 36 months
  Overall remission rate, according to Lugano 2014 criteria.

OTHER OUTCOMES:
PFS | Up to 36 months
  Progression-free survival
OS | Up to 36 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No